CLINICAL TRIAL: NCT06680531
Title: A Clinical Study to Evaluate the Drug Interaction Between YZJ-1139 Tablets and Escitalopram Oxalate Tablets
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: YZJ-1139-1-14
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Insomnia; Central Nervous System
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Drug interaction
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: YZJ-1139 tablets; Drug: Escitalopram oxalate tablets; Drug: YZJ-1139 simulated tablets
- Group B (Placebo Comparator)
  Interventions: Drug: Escitalopram oxalate tablets; Drug: YZJ-1139 simulated tablets

INTERVENTIONS:
Drug: YZJ-1139 tablets — YZJ-1139 tablets are administered orally single dose
  Arms: Group A
Drug: Escitalopram oxalate tablets — •oral tablet, QD
Drug: YZJ-1139 simulated tablets — oral tablet, QD

SUMMARY:
Primary Objective：

1) To evaluate the pharmacodynamic interaction between YZJ-1139 tablets and Escitalopram oxalate tablets in healthy subjects; 2) To evaluate the pharmacokinetic interaction between YZJ-1139 tablets and Escitalopram oxalate tablets in healthy subjects; To observe the safety of YZJ-1139 tablets taken together with Escitalopram oxalate tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 45 years (inclusive);
2. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 28.0 kg/m2 (inclusive);
3. Subjects with normal physical examination, vital signs, 12-lead ECG and laboratory tests results or abnormal but no clinical significance;
4. Subjects who are in good health and have no history of serious or chronic diseases such as respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system;
5. Subjects of childbearing potential (including partners) have no family planning or donate sperm/eggs from 2 weeks before screening to 3 months after dosing, and voluntarily take appropriate contraceptive measures;
6. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.

Exclusion Criteria:

1. Allergic constitution, such as those with a known history of allergies to two or more drugs or foods, or those with a history of allergies to experimental drugs or excipients;
2. Subjects with difficulty swallowing tablets and special dietary requirements who cannot accept a unified diet;
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting;
4. Subjects who have undergone surgery within 30 days prior to screening, or plan to undergo surgery during the study;
5. Individuals with a history of paroxysmal sleep disorder, obstructive sleep apnea, complex sleep behavior (such as dream walking, driving in dreams, etc.), severe unconscious hypoglycemia, stroke, epilepsy, and other psychiatric disorders (including anxiety, depression, etc.), convulsive diseases, and sudden onset of illness;
6. Known to have QT prolongation or congenital QT syndrome or screening period electrocardiogram showed QTc interval (QTcF)>450 msec in males and>470 msec in females（QTcF= QT/(RR^0.33)）;
7. Those who are positive in any index screening of hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum-specific antibody, and human immunodeficiency virus antibody;
8. Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening;
9. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, alcohol or 150 mL of wine), or who cannot stop using any alcohol products during the study, or whose alcohol breath test result > 0.0 mg/100 mL;
10. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, received blood transfusions or used blood products, planned to donate blood during the trial period or within 1 month after the end of the trial;
11. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup ≈ 250 mL) daily during the 3 months before screening;
12. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study;
13. Subjects who have participated in any clinical trial and have used clinical trial drugs or medical device within 3 months prior to screening, or plan to participate in other clinical trials during the study;
14. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study;
15. Subjects who have used any drugs that inhibit or induce hepatic metabolism of drugs within 30 days prior to admission (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines);
16. Subjects who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, and Chinese herbal medicines within 14 days before administration;
17. Subjects who have consumed grapefruit, pomelo, pitaya, mango and other fruits or related products affecting metabolic enzymes within 14 days before administration;
18. Subjects who have ingested caffeine-rich or xanthine-rich beverages or foods (such as coffee, strong tea, chocolate, cola, etc.) within 48 h before administration;
19. Lactating women, or women who test positive for pregnancy;
20. Subjects with acute illness from screening period to pre-dose;
21. Those who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
saccade eye movement test | From Day 1 to Day 11
  Saccadic eye movements were evaluated by using a computer-based electronystagmography system.To assess the change in scores for escitalopram oxalate tablets combined with YZJ-1139 tablets relative to YZJ-1139 tablets simulant and YZJ-1139 tablets.
body swing test | From Day 1 to Day 11
  Body swing test was measured with an apparatus, which integrates the amplitude of unidirectional body sway. To assess the change in scores for escitalopram oxalate tablets combined with YZJ-1139 tablets relative to YZJ-1139 tablets simulant and YZJ-1139 tablets.
selective reaction time test | From Day 1 to Day 11
  Subjects selected buttons in different directions according to Chinese character prompts on a computer screen,assess the change in scores for escitalopram oxalate tablets combined with YZJ-1139 tablets relative to YZJ-1139 tablets simulant and YZJ-1139 tablets.
number symbol conversion test | From Day 1 to Day 11
  Subjects click the corresponding number according to the corresponding relationship between the given symbol and the number. To assess the change in scores for escitalopram oxalate tablets combined with YZJ-1139 tablets relative to YZJ-1139 tablets simulant and YZJ-1139 tablets.
word memory test | From Day 1 to Day 11
  Subjects recall presented words at specific times.To assess the change in scores for escitalopram oxalate tablets combined with YZJ-1139 tablets relative to YZJ-1139 tablets simulant and YZJ-1139 tablets.
Maximum Observed Plasma Concentration (Cmax) of YZJ-1139 | From Day 1 to Day 11
  Cmax is defined as the maximum concentration of drug.
Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC0-t) of YZJ-1139 | From Day 1 to Day 11
  AUC0-t is defined as the concentration of drug from time zero to the last observable concentration.
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of YZJ-1139 | From Day 1 to Day 11
  AUC0-∞ is defined as the concentration of drug extrapolated to infinite time.
Time of Maximum Observed Plasma Concentration (Tmax) of Entrectinib | From Day 1 to Day 11
  Tmax is defined as the time (observed time point) of Cmax.
Apparent Terminal Elimination Half-life (t1/2) of Entrectinib | From Day 1 to Day 11
Apparent Oral Clearance (CL/F) of Entrectinib | From Day 1 to Day 11
  CL/F is defined as the apparent oral clearance following administration of the drug.
The Apparent Volume of Distribution (Vz/F) of Entrectinib | From Day 1 to Day 11
  Vz/F is defined as the apparent volume of distribution of the drug.
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, China